CLINICAL TRIAL: NCT03552666
Title: A Randomized, Examiner-blind Comparator-controlled Crossover Bioequivalence Study on Vitamin D in Healthy Adults
Brief Title: Clinical Study on the Bioequivalence of Vitamin D in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ST-7639N9
Record Dates: First submitted 2018-05-02; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Bioequivalence of Vitamin D in Healthy Adults
Keywords: Vitamin D
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized, examiner-blind, comparator-controlled crossover study
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitafusion Extra Strength Vitamin D3 Gummy (Experimental): A single oral dose of gummy vitamin D3 to monitor Vitamin D blood levels
  Interventions: Dietary Supplement: vitamin D3
- Nature Made Vitamin D3 Tablet (Active Comparator): A single oral dose of tablet vitamin D3 to monitor Vitamin D blood levels
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3

SUMMARY:
The objective of this clinical study is to evaluate and compare the bioequivalence between a single oral dose of vitamin D3 gummy vitamin versus vitamin D3 tablet in healthy adults.

DETAILED DESCRIPTION:
The investigators hypothesize that the gummy and tablet preparations of vitamin D3 supplement will be biologically equivalent, as defined by the absence of a statistically significant difference in bioavailability measured as blood levels of vitamin D3 after administration of the same oral dose of vitamin D3 as gummy and tablet supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Females not of childbearing potential (i.e., hysterectomy, oophorectomy, bilateral tubal ligation or postmenopausal) or females of childbearing potential that agree to use a medically approved method of birth control such as hormonal contraceptives, double-barrier, non-hormonal intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s) and/or vasectomy of partner
* BMI 18.5 to 29.9 kg/m2
* Agrees to maintain current level of physical activity throughout the study
* Agrees to wear sunblock of at least SPF 45 during the study and not to have excessive sun exposure (no more than 1 hour without sunblock)

Exclusion Criteria:

* Women who are pregnant to be determined by UPT (urine pregnancy test), breastfeeding, or planning to become pregnant during the course of the study
* Duodenal ulcer or gastric ulcer, gastritis, hiatus hernia, or GERD within the past 3 months
* Significant gastrointestinal disease, history of malabsorption, or history of irritable bowel syndrome and related disorders
* Unstable medical conditions as determined by the principal investigator
* Clinically significant abnormal laboratory results on CBC or BMP at screening
* Cancer chemotherapy/radiation treatment within the 3 months prior to enrollment
* Metabolic disease
* History of kidney stones
* Use of prescription or over the counter products known to interact with vitamin D within 72 hours of randomization and during the trial such as aspirin and NSAIDs, aluminum, iron and proton pump inhibitors
* Use of acute over the counter medication within 72 hours of test product dosing
* Smokers
* Consumption of more than 2 alcoholic drinks per day
* Drug abuse within the past year
* Use of medicinal marijuana
* Immunocompromised individuals such as individuals that have undergone organ transplantation or individuals diagnosed with human immunodeficiency virus (HIV)
* Individuals who have planned surgery during the course of the trial
* Use of St. John's wort in the last 30 days before randomization and during the study
* Use of vitamin D, multivitamins containing vitamin D, foods or beverages fortified with vitamin D and other natural healthy products containing vitamin D, or consumption of grapefruit/ grapefruit juice within 14 days of randomization and during the study
* Use of anticoagulants , barbiturates, tetracycline antibiotics, beta-blockers, cyclosporine, prednisone, tricyclic antidepressants, diuretics and nitrate medications
* History of blood/bleeding disorders
* Anemia of any etiology defined as hemoglobin < 140 g/L for males and < 123 g/L for females
* Blood donation in the past 3 months, or individuals planning to donate blood during the study or within 30 days of completion of study
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to any ingredient in supplements provided during the study
* Individuals who are cognitively impaired and/or who are unable to give informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-26 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Mean Absorption | baseline, 3, 6, 10, 24 and 48 hours
  A comparison of mean absorption of the two vitamin formulations (gummy vs. tablet)

SECONDARY OUTCOMES:
Absorption Rate | 0 to 48 hours
  A comparison of absorption rate across the two vitamin formulations (gummy vs. tablet)

CONTACTS AND LOCATIONS:
Locations (1):
- Church & Dwight Co., Inc., Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No